CLINICAL TRIAL: NCT03120520
Title: A Randomized, Double-blind, Placebo-controlled, 3 Dose Level, Parallel Group Study of the Efficacy and Safety of Plecanatide in Adolescents 12 to < 18 Years of Age With Chronic Idiopathic Constipation (CIC)
Brief Title: An Efficacy and Safety Study of Plecanatide in Adolescents 12 to <18 Years of Age With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP304202-13
Record Dates: First submitted 2017-04-18; First posted 2017-04-19 (Actual); Results first posted 2019-09-19 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-08

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Plecanatide 0.5 mg (Experimental): Taken orally once daily in the morning for 8 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 1.0 mg (Experimental): Taken orally once daily in the morning for 8 weeks
  Interventions: Drug: Plecanatide
- Plecanatide 1.5 mg (Experimental): Taken orally once daily in the morning for 8 weeks
  Interventions: Drug: Plecanatide
- Matching placebo (Placebo Comparator): Taken orally once daily in the morning for 8 weeks
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Plecanatide
  Other Names: Trulance
  Arms: Plecanatide 0.5 mg; Plecanatide 1.0 mg; Plecanatide 1.5 mg
Drug: Matching placebo
  Other Names: No other names
  Arms: Matching placebo

SUMMARY:
This is a study of efficacy and safety of Plecanatide in pediatric subjects aged 12 to < 18 years diagnosed with Chronic Idiopathic Constipation.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate efficacy, safety, and pharmacokinetics (PK) of oral Plecanatide 0.5, 1.0 and 1.5 mg tablets dosed once a day as compared to matching placebo, when administered for 8 weeks in adolescents with chronic idiopathic constipation.

This study will consist of a 4-week screening period, 8 weeks of treatment, and a 2-week follow-up. The study will assess the effects of Plecanatide on bowel movement frequency and other clinical features of CIC.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female adolescents 12 to less than 18 years of age.
2. Diagnosed with CIC based on the Rome III criteria for child/adolescent functional constipation (Appendix A).
3. Patient is able to voluntarily provide written, signed, and dated (personally and via a legally authorized representative [LAR]) assent/informed consent as applicable to participate in the study.
4. Subject's parent/LAR demonstrates an understanding, ability, and willingness to fully comply with study procedures (e.g., accept venipuncture, willing and able to swallow tablets, accept urine drug screen for opiates) and restrictions.

Key Exclusion Criteria:

1. The patient has a mental age <4 years in the investigator's opinion.
2. The patient has previously been diagnosed with anorectal malformations, neurological deficits, or anatomical anomalies that would constitute a predisposition to constipation.
3. The patient currently requires iron supplements, amitriptyline, or other tricyclic antidepressants for depression, opioid-containing medications or compounds for pain, or has other conditions that require medications known to cause constipation. A patient with an onset of constipation prior to the use of these medications and who has been on a stable dose for at least 8 weeks prior to Screening might be considered eligible for this study if the investigator deems these medications do not significantly contribute to the patient's constipation. Screening of these patients needs to be approved by the medical monitor and the sponsor.
4. The patient, if female of childbearing potential (defined as postmenarche), does not agree to practice 1 of the following medically acceptable methods of birth control throughout the study:

   * Hormonal methods such as oral, implantable, injectable, vaginal ring, or transdermal contraceptives for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before study drug administration.
   * Total abstinence from sexual intercourse since the last menses before study drug administration.
   * Intrauterine device.
   * Double barrier method (condoms, sponge, or diaphragm with spermicidal jellies or cream.
5. The patient follows a diet not considered normal by the investigator for the patient's age, relative to variety of food, caloric content, and quantity. The patient must have been on a stable diet for at least 30 days weeks prior to Screening.
6. The patient's mobility or normal exercise tolerance is compromised in the investigator's opinion.
7. The patient has a history of an eating disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Synergy Research Site, Foley, Alabama
  - Synergy Research Site, Jonesboro, Arkansas
  - Synergy Research Site, Cerritos, California
  - Synergy Research Site, Corona, California
  - Synergy Research Site, Downey, California
  - Synergy Research Site, Huntington Beach, California
  - Synergy Research Site, Sacramento, California
  - Synergy Research Site, Ventura, California
  - Synergy Research Site, Wilmington, Delaware
  - Synergy Research Site, DeLand, Florida
  - Synergy Research Site, Doral, Florida
  - Synergy Research Site, Hialeah, Florida
  - Synergy Research Site, Miami, Florida
  - Synergy Research Site, Orlando, Florida
  - Synergy Research Site, Tampa, Florida
  - Synergy Research Site, Snellville, Georgia
  - Synergy Research Site, Thomaston, Georgia
  - Synergy Research Site, Idaho Falls, Idaho
  - Synergy Research Site, Meridian, Idaho
  - Synergy Research Site, Nicholasville, Kentucky
  - Synergy Research Site, Crowley, Louisiana
  - Synergy Research Site, Bellevue, Nebraska
  - Synergy Research Site, Omaha, Nebraska
  - Synergy Research Site, Fayetteville, North Carolina
  - Synergy Research Site, Cincinnati, Ohio
  - Synergy Research Site, Columbus, Ohio
  - Synergy Research Site, Dayton, Ohio
  - Synergy Research Site, Gresham, Oregon
  - Synergy Research Site, Jackson, Tennessee
  - Synergy Research Site, Kingsport, Tennessee
  - Synergy Research Site, Memphis, Tennessee
  - Synergy Research Site, Corpus Christi, Texas
  - Synergy Research Site, Houston, Texas
  - Synergy Research Site, McAllen, Texas
  - Synergy Research Site, San Antonio, Texas
  - Synergy Research Site, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Matching Placebo: Taken orally once daily in the morning for 8 weeks
  Matching placebo
- Plecanatide 0.5 mg; Plecanatide 1.0 mg; Plecanatide 1.5 mg: Taken orally once daily in the morning for 8 weeks
  Plecanatide
Period: Overall Study
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
Started | 31 | 31 | 30 | 32
Completed | 27 | 27 | 26 | 29
Not Completed | 4 | 4 | 4 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 2
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg | Total
Number analyzed (Participants) | 31 | 31 | 30 | 32 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.61) | 15.1 (1.48) | 14.5 (1.89) | 14.6 (1.52) | 14.7 (1.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 17 | 18 | 69
  Male | 14 | 14 | 13 | 14 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 23 | 27 | 92
  Not Hispanic or Latino | 10 | 10 | 7 | 5 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 3 | 2 | 16
  White | 24 | 24 | 27 | 29 | 104
  More than one race | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 30 | 32 | 124
Baseline Stool Consistency [Mean (Standard Deviation); unit: units on a scale] — Stool consistency was assessed via the 7-point (1-7) Bristol Stool Form Scale (BSFS) and recorded in the Bowel Movement (BM) and Symptom Diaries. Types were 1) separate hard lumps, like nuts (hard to pass); 2) sausage-shaped but lumpy; 3) like a sausage but with cracks on its surface; 4) like a sausage or snake, smooth and soft; 5) soft blobs with clear-cut edges (passed easily); 6) fluffy pieces with ragged edges, a mushy stool; 7) watery, no solid pieces, entirely liquid. Baseline is the mean of the BSFS scores recorded during the 2-week baseline diary period prior to the first dose of drug.
  units on a scale | 2.17 (0.932) | 2.0 (1.190) | 2.08 (.899) | 2.29 (1.298) | 2.13 (1.140)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Overall Responders
Description: An Overall Responder is a participant who was a Spontaneous Bowel Movement (SBM) responder for the last 2 weeks of the Treatment Period. An SBM responder is defined as a participant who had >3 SBMs per week. SBM was defined as a bowel movement that occurs in the absence of laxative use within the preceding 24 hours. Participants missing with respect to the outcome measure were scored as non-responders.
Time Frame: 8 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
Number analyzed (Participants) | 31 | 31 | 30 | 32
Participants | 7 | 10 | 12 | 7

2. Secondary Outcome: Change From Baseline in Weekly Average Stool Consistency Bristol Stool Form Scale (BSFS) Score
Description: Stool consistency was assessed via the 7-point (1-7) Bristol Stool Form Scale (BSFS) and recorded in the bowel movement (BM) and Symptom Diaries. Lower numbers represent more formed stools; higher numbers represent less formed stools. The weekly mean BSFS score per patient = (total of all BSFS scores reported for a corresponding Spontaneous Bowel Movement (SBM) per time period)/n, where n = number of SBMs scored during the time period. Baseline was the mean BSFS score recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. BSFS types were 1) separate hard lumps, like nuts (hard to pass); 2) sausage-shaped but lumpy; 3) like a sausage but with cracks on its surface; 4) like a sausage or snake, smooth and soft; 5) soft blobs with clear-cut edges (passed easily); 6) fluffy pieces with ragged edges, a mushy stool; 7) watery, no solid pieces, entirely liquid.
Time Frame: 8 weeks
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
Number analyzed (Participants) | 31 | 31 | 30 | 32
units on a scale | 0.98 (0.209) | 1.09 (0.209) | 1.22 (0.205) | 1.06 (0.191)

3. Secondary Outcome: Change From Baseline in the Weekly Rate of Spontaneous Bowel Movements (SBM)
Description: The weekly Spontaneous Bowel Movement (SBM) totals were derived from the daily diary entries reported during the Treatment Period in the Bowel Movement (BM) and symptom diaries. Baseline was the mean number of SBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. SBM is defined as a bowel movement that occurs in the absence of laxative use within the preceding 24 hours
Time Frame: 8 weeks
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: Weekly SBMs
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
Number analyzed (Participants) | 31 | 31 | 30 | 32
Weekly SBMs | 1.44 (0.332) | 1.97 (0.339) | 2.06 (0.343) | 2.05 (0.328)

4. Secondary Outcome: Change From Baseline in the Weekly Rate of Complete Spontaneous Bowel Movements (CSBM)
Description: The weekly Complete Spontaneous Bowel Movement (CSBM) totals are derived from the daily diary entries reported during the Treatment Period in the Bowel Movement (BM) and symptom diaries. Baseline is the mean number of CSBMs recorded during the 2-week baseline diary assessment period prior to the first dose of study drug. Spontaneous Bowel Movement (SBM) was defined as a bowel movement that occurs in the absence of laxative use within the preceding 24 hours. CSBM was defined as a spontaneous bowel movement with the sense of complete evacuation.
Time Frame: 8 weeks
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: Weekly CSBMs
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
Number analyzed (Participants) | 31 | 31 | 30 | 32
Weekly CSBMs | 1.30 (0.344) | 1.71 (0.348) | 1.83 (0.354) | 2.11 (0.340)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Matching Placebo | Plecanatide 0.5 mg | Plecanatide 1.0 mg | Plecanatide 1.5 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 4/31 | 7/31 | 4/30 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Matching Placebo (N=31) | Plecanatide 0.5 mg (N=31) | Plecanatide 1.0 mg (N=30) | Plecanatide 1.5 mg (N=32)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 1
Acute Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Infectious Mononucleosis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal Discomfort (General disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Gilbert's syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1
Decreased apetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact Sponsor for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT03120520/Prot_SAP_000.pdf